CLINICAL TRIAL: NCT01214824
Title: Use of the FreeStyle Navigator Continuous Glucose Monitoring System to Enhance Education and Glycaemic Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Diabetes Care (Industry)
Collaborators: Liverpool University Hospitals NHS Foundation Trust (Other Government); National Heatlh Service Ayrshire and Arran (Other Government); NHS Lothian (Other Government); National Health Service, United Kingdom (Other Government); Cardiff and Vale University Health Board (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADC-PMR-NAV-09005
Record Dates: First submitted 2010-10-04; First posted 2010-10-05 (Estimated); Results first posted 2013-06-06 (Estimated); Last update posted 2013-07-02 (Estimated); Status verified 2013-06

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes; Continuous Glucose Monitoring
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: FreeStyle Navigator Continuous Glucose Monitoring System — Six x 5 day wears of the continuous glucose monitoring device. Two of the 6 wears will be using a masked device (1 at the start and 1 at the end of the study).

SUMMARY:
To demonstrate that in patients with persistent poorly controlled diabetes, short/intermittent use of continuous glucose monitoring can driver better longer-term glycaemic control and HbA1c.

DETAILED DESCRIPTION:
Study Overview This is a multi-centre pilot study across 6 study sites, recruiting 50 subjects. Each subject will use a FreeStyle Navigator Continuous Glucose Monitor for a period of 20 days at the start of the study, after which their Healthcare Professionals (HCPs) may recommend changes to their glucose management based on the continuous glucose monitoring(CGM) data. Subjects will then return to self-managing their diabetes with a blood glucose meter. After 2 months, subjects will use the FreeStyle Navigator for a further 5 days and review their results and glucose management with their HCPs. Subjects will again return to self-managing their diabetes with a blood glucose meter until the end of the study, when the last FreeStyle Navigator 5 day wear is completed and HbA1c and measures of glycaemic variability are recorded.

ELIGIBILITY:
Inclusion Criteria:

* Subject with Type 1 or Type 2 diabetes requiring Multiple Daily Injections (MDI) (for >1yr)
* Age 18-65 years
* HbA1c above 8.0% for previous 2 HbA1c tests; the last HbA1c result being obtained within 3 months prior to enrolment
* Completed a structured education programme meeting NICE criteria between 6 to 24 months prior to enrolment.
* Testing Blood Glucose ≥ 4 times a day for previous 12 months

Exclusion Criteria:

* Subject is currently on an insulin pump.
* Subject has known allergy to medical grade adhesives
* Subject has concomitant disease that influences metabolic control
* Subject is participating in another study of a glucose monitoring device / drug that could affect glucose measurements / management
* Subject is currently using another continuous glucose monitoring device or has previously used real-time continuous glucose monitoring.
* Subject is receiving peritoneal dialysis solutions containing icodextrin
* Subject is pregnant / planning to become pregnant during study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-11; Primary Completion 2012-02 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jiten Vora, MRCP, Principal Investigator — The Royal Liverpool and Broadgreen University Hospitals NHS Trust
Locations (5):
- United Kingdom (5):
  - Ayr Hospital, Ayr, Ayrshire
  - The Royal Liverpool University Hospital, Liverpool, Cheshire
  - University Hospital Aintree, Liverpool, Cheshire
  - Glan Clywd Hospital, Rhyl, Denbighshire
  - St. John's Hospital, Livingston, Edinburgh

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with type 1 or type 2 diabetes on Multiple Daily Injection(MDI)of insulin(3 or more injections per day)with an HbA1c of 8% or more for their last two tests were recruited at five sites across the United Kingdom. The target enrolment was 50 subjects, with the aim of completing the study with 40 subjects for statistical analysis.
Groups:
- Intervention Group: Participants using the FreeStyle Navigator System Intermittently. At the start and end of the study subjects wore the FreeStyle Navigator masked (without seeing continuous glucose results) for 5 days (1 sensor wear). During the study subjects used the FreeStyle Navigator fully functional (unmasked) for 2 periods. The first unmasked phase was for 2 weeks (3 sensor wears) following the baseline masked wear. The second unmasked phase was a 5 day wear at 3 months. After each unmasked phase the HCP reviewed results with the subject and changes to insulin regimen were recommended as required. For the remainder of the study a standard blood glucose meter was used for diabetes management.
Period: Overall Study
Arm/Group | Intervention Group
Started | 32
Completed | 29
Not Completed | 3

BASELINE CHARACTERISTICS:
Groups:
- Intervention Group: Participants using the FreeStyle Navigator System Intermittently
Arm/Group | Intervention Group
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 32
  >=65 years | 0
Age Continuous [Mean (Full Range); unit: years] | 42.5 [18 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 9
Body Mass Index (BMI) [Mean (Full Range); unit: kg/m^2] | 26.3 [19.6 to 37.0]
Weight [Mean (Full Range); unit: Kg] | 73.7 [49 to 115]
Years since diagnosis [Mean (Full Range); unit: Years] | 17.6 [0.7 to 48]
Daily Total Insulin Dosage-Basal [Mean (Full Range); unit: Units] | 24.9 [0 to 62]
Daily Total Insulin Dosage-Bolus [Mean (Full Range); unit: Units] | 28.0 [10 to 60]
Number of injections per day [Mean (Full Range); unit: Injections] | 4.1 [3 to 6]
Number of blood glucose measurements per day [Mean (Full Range); unit: Tests] | 4.5 [4 to 10]
HbA1c [Mean (Full Range); unit: %] | 9.3 [8.0 to 13.2]

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1C From Baseline to 6 Months
Description: HbA1c at baseline HbA1c at 6 months Change in HbA1c(%)(6 months - baseline)
Time Frame: Baseline and 6 months
Population: Intention to treat analysis
Measure: Mean (Standard Deviation); unit: HbA1c %
Arm/Group | Intervention Group
Number analyzed (Participants) | 32
HbA1c %
  Baseline | 9.3 (1.3) [-0.8 to 0.0]
  6 months | 9.1 (1.3)
Statistical Analysis 1: Comparison: Intervention Group; Comparison is HbA1c at 6 months versus Baseline; Test type: Superiority or Other; p = 0.014, Wilcoxon signed rank test; Median Difference (Final Values) = -0.3

2. Secondary Outcome: Number of Subjects Who Had Reduction in HbA1c of > or = 0.5%
Description: Number of subjects with a HbA1c reduction greater than or equal to 0.5% and 95% confidence interval from visit 1 (baseline) to visit 7 (6 months).
Time Frame: Baseline and 6 months
Population: Intention to treat analysis
Measure: Number; unit: participants
Arm/Group | Intervention Group
Number analyzed (Participants) | 32
participants | 14

3. Secondary Outcome: Proportion of Time in Hypoglycaemia (<3.9 mmol/L)- Masked
Description: Proportion of time (hours per day) in hypoglycaemia (<3.9 mmol/L) for the masked phase. There were two masked phases in the study, one 5 day wear at baseline and one 5 day wear at 6 months. During masked wear subject were not able to see continuous glucose data from the device.
Time Frame: Baseline & 6 months
Population: Analysis per protocol
Measure: Mean (Standard Deviation); unit: Hours per day
Arm/Group | Intervention Group
Number analyzed (Participants) | 28
Hours per day
  Time in hypoglycaemia (<3.9mmol/L)-masked phase 1 | 0.93 (0.84)
  Time in hypoglycaemia (<3.9mmol/L)-masked phase 2 | 1.06 (1.02)
Statistical Analysis 1: Comparison: Intervention Group; Comparison is masked phase 2 versus masked phase 1; Test type: Superiority or Other; p = 0.5304, Paired t-test

4. Secondary Outcome: Proportion of Time in Hypoglycaemia (<3.9mmol/L)-Unmasked
Description: Proportion of time (hours per day) in hypoglycaemia (<3.9mmol/L) for the unmasked phase
Time Frame: 2 weeks following baseline & 3 months
Population: Analysis per protocol 31 participants analysed in the unmasked phase 1 28 participants analysed in the unmasked phase 2
Measure: Mean (Standard Deviation); unit: Hours per day
Arm/Group | Intervention Group
Number analyzed (Participants) | 31
Hours per day
  Time in hypoglycaemia(3.9mmol/L)unmasked phase 1 | 0.60 (0.47)
  Time in hypoglycaemia(3.9mmol/L)unmasked phase 2 | 0.49 (0.55)

ADVERSE EVENTS:
Arm/Group | Intervention Group
Serious Adverse Events (participants affected / at risk) | 3/32
Other Adverse Events (participants affected / at risk) | 3/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Group (N=32)
Right iliac fossa pain (General disorders) | 1 (1) — Not device related, not related to study procedure, severity - moderate
Unresolving Paronychia (Skin and subcutaneous tissue disorders) | 1 (1) — Not device related, not related to study procedure, severity - moderate
Viral Meningitis (Infections and infestations) | 1 (1) — Not device related, not related to study procedure, severity - moderate
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Group (N=32)
Infection (Infections and infestations) | 1 (1) — Not device related, not related to study procedure, severity - mild
Abdominal pain (muscle strain) (Musculoskeletal and connective tissue disorders) | 1 (1) — Not device related, not related to study procedure, severity - moderate
Broken toe (Musculoskeletal and connective tissue disorders) | 1 (1) — Not device related, not related to study procedure, severity - moderate

LIMITATIONS AND CAVEATS:
After an enrolment review recruitment was ceased on 02 Sep 11 with only 32/50 enrolled subjects. The screening/recruitment phase had been 12 weeks but was significantly extended. Only 7/32 subjects had completed 6 month HbA1c when recruitment ceased.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days